CLINICAL TRIAL: NCT04313699
Title: Diagnosis and Treatment of Non-communicable Diseases and Geriatric Syndromes in the HIV Aging Population in Sub-Saharan Africa
Brief Title: Geriatric HIV Cohort in Sub Sahara Africa
Acronym: HASA
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Makerere University (Other)
Responsible Party: Sponsor
Other Study IDs: TMA2017GSF-1936
Record Dates: First submitted 2020-03-04; First posted 2020-03-18 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: HIV Infections; Non Communicable Diseases; Aging
MeSH Terms: conditions — HIV Infections; Noncommunicable Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Packed cells Plasma Serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Antiretroviral treatment — The cohort will recruit HIV infected participants who are on antiretroviral treatment
  Other Names: Assessment of non communicable diseases and geriatric syndromes

SUMMARY:
The overall goal of the proposal is to improve capacity for detection and management of non-communicable diseases and geriatric syndromes in the aging HIV population in sub-Saharan Africa

DETAILED DESCRIPTION:
The establishment and scale up of solid and sustainable HIV programs in sub-Saharan Africa (SSA) has led to a reduction in mortality and morbidity from HIV related opportunistic infections and some HIV related cancers. This improved survival has resulted in two phenomena: the first is the surfacing of non-communicable diseases (NCDs) in the HIV population, especially in those on long-term ART, and the second is increased longevity leading to increasing numbers of elderly HIV infected individuals

ELIGIBILITY:
Inclusion Criteria:

Age 60 years and above

* Evidence of a personally signed and dated informed consent document indicating that the subject (or a legal representative) has been informed of all pertinent aspects of the study.
* Subjects who are willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

* Any clinical (physical and psychiatric) condition which prevents the patients to participate safely in the study procedures according to the judgments of a physician.
* Subjects already enrolled in experimental clinical trial.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients 60 years and above at IDI are referred to the elderly specialist clinic, which is run once a week by a physician, therefore study participants will be identified from this clinic. Enrolment into the Geriatric cohort will be offered to all patients 60 years and above attending attending their monthly routine clinic visit at the elderly specialist clinic will be approached by the study staff, will be given detailed information and be asked if they are willing to participate.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-07-01 (Estimated); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in proportion of participants with any non communicable disease | Enrollment, year 1, year 2
  Proportion with any non communicable disease (including hypertension, cardio vascular disease, respiratory disease, renal disease, non HIV related cancers, frailty)
Change in Quality of life | Enrollment, year 1, year 2
  Quality of life measured using the WHO Quality of life for elderly (WHOQOL-OLD)

SECONDARY OUTCOMES:
Change in proportion of patients with polypharmacy monitoring | Enrollment, year 1, year 2
  Polypharmacy defined as 5 or more drugs beyond antiretroviral drugs, used in the same individuals for more than 4 weeks. Information of polypharmacy will be collected by the clinic files and self reported by the participants
Change in Nutritional status assessed by Mini Nutritional Assessments (MNA) | Enrollment, year 1, year 2
  Nutrition screening and assessment to identify geriatric patients age who are malnourished or at risk of malnutrition.
Change in proportion of patients with history of falls | Enrollment, year 1, year 2
  Occurrence of falls measured with the History of Falls questionnaire
Change in proportion of patients with urinary incontinence measured by ICIQ-UI Short | Enrollment, year 1, year 2
  Presence of urinary incontinence measured with the Internal Consultation on Incontinence Questionnaire
Change in proportion of patients with depression | Enrollment, year 1, year 2
  Depression measurement using the People Health Questionnaire-9 (scale 0-30, higher: worse)
Change in proportion of patients with disability | Enrollment, year 1, year 2
  Assessment of the Instrumental Activities of Daily Living (score 0-8, higher: better)
Change in proportion of patients with cognitive deficit | Enrollment, year 1, year 2
  Screening using Montreal Cognitive Assessment (score 0-30; higher: better)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Castelnuovo, PhD, Principal Investigator — Infectious Diseases Institute (IDI)

IPD SHARING:
Plan to Share IPD: Yes
At the end of the project the dataset generated from the study will be made available as per the EDCTP Horizon 2020 guidelines. These data will be de-identified prior to sharing widely. The data will be shared in form an excel CSV spreadsheet that will be shared by the PI once the necessary approvals are met. We currently do not have a repository for the data, however at the time of publishing in Open Access Journals, the data will be made available
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: 2025-2030
Access Criteria: Approval from the PI